CLINICAL TRIAL: NCT02474992
Title: The Kanyakla Study: a Microclinic Social Network Intervention for Promoting Engagement and Retention in HIV Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Organic Health Response (Other); Microclinic International (Other); Kenya Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OHR006
Record Dates: First submitted 2015-06-16; First posted 2015-06-18 (Estimated); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: HIV
Keywords: HIV; Social network; Social support; Disclosure; Stigma; Kenya
MeSH Terms: conditions — Social Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): This arm is eligible for participation in the Microclinic intervention, a social network-based educational program.
  Interventions: Behavioral: Microclinic
- Comparison (No Intervention): This arm is not eligible for participation in the intervention during the first twelve months of the study. Following collection of the primary study endpoints, this arm will also be invited to participate in a Microclinic group. Participants in this arm will still have access to standard HIV care at the facility of their choice. At time of recruitment into the study, prior to randomization, all eligible participants will be counseled on the importance of returning to their clinic for ongoing HIV care.

INTERVENTIONS:
Behavioral: Microclinic — Individuals randomized to this arm will be invited to recruit members of their social network to form a health team, or microclinic. These groups will proceed through a discussion-based health education curriculum led by local community health workers. Topics will include HIV biology, medications, the importance of social support, and community outreach for reducing HIV stigma. The curriculum will conclude with an opportunity for all group members to disclose their HIV status to one another.
  Other Names: Kanyakla
  Arms: Intervention

SUMMARY:
The purpose of this randomized controlled trial is to compare a social network-based behavioral intervention known as microclinics to standard HIV clinical care alone in helping patients receiving HIV care on Mfangano, Remba and Ringiti Islands, Kenya remain adherent to clinic appointments. The study is designed to evaluate the effectiveness of microclinics on reducing gaps in clinical care, HIV viral load and HIV-related stigma, compared to standard HIV clinical care alone. By doing this research study, the investigators hope to learn whether microclinics are a useful social strategy for improving delivery of HIV treatment in rural Kenya.

ELIGIBILITY:
Inclusion Criteria:

* Must be currently receiving combination antiretroviral therapy (cART) or co-trimoxozole prophylaxis from one of the eligible study clinics:

  * Is currently in care at study baseline, defined as having ≥1 medical care visit to receive medications (cART or prophylaxis) during the six months preceeding initiation of study enrollment, OR
  * Initiates pre-ART or ART care for the first time at a study clinic during the six month study recruitment period, OR
  * Transfers from a clinic outside the study area and receives pre-ART or ART care for the first time from a study clinic during the six month recruitment period
* Participants become eligible for study inclusion on the 4th day following a missed clinic appointment, provided the patient has not transferred care to another clinic prior to the 4th day, moved outside the study area or died. Participants who miss a study visit by >3 days but return to clinic before recruitment takes place are still eligible for study enrollment. Missed visits must have occurred within the previous 90 days at the time of eligibility assessment to meet this inclusion criteria.
* Must currently reside on Mfangano, Remba or Ringiti Island.
* Must be conversant with one of the commonly spoken languages within the study area (i.e. DhoLuo, Swahili or English; prior experience indicates that this represents >99% of the adult population).
* Must be ≥18 years of age as of the date of study eligibility.

Exclusion Criteria:

* Eligible participants who reside in the Mfangano East sub-location will be excluded from participation in this study. Many of these patients have already participated in the microclinic intervention as part of the Mfangano Island Healthy Network Impact Study.
* Participants planning on moving permanently out of the study area within the next six months will be excluded.
* Participants who, should they be randomized to the intervention arm, would be unwilling to participate in a microclinic will be excluded from study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2016-01; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Disengagement from care | 12 months
  Incidence of 90-day absence from care following a missed appointment
Disengagement from care | 12 months
  Proportion of time eligible for HIV care that patient is adherent to clinic appointment schedules. Calculated by subtracting the sum of all gaps in care from the total time eligible for care, and dividing by total time eligible for care. Gaps in care are defined as the number of days between a missed appointment and subsequent return to any clinic in the study area to access HIV care.

SECONDARY OUTCOMES:
Virologic suppression | 12 months
  Proportion of patients who are virologically suppressed 12 months after randomization
HIV-related stigma | 12 months
  Reduction in stigma as compared to baseline, measured by the Earnshaw HIV Stigma Framework
Re-engagement in care | 12 months
  Incidence of re-engagement in care following missed visit at time of study enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Craig R Cohen, MD, MPH, Principal Investigator — University of California, San Francisco; Elizabeth A Bukusi, MBChB, M.Med, PhD, Principal Investigator — Kenya Medical Research Institute; Matthew D Hickey, MD, Principal Investigator — University of California, San Francisco; Charles R Salmen, MD, MPhil, Principal Investigator — Organic Health Response
Locations (1):
- Ekialo Kiona Center, Mfangano Island, Homa Bay County, Kenya

REFERENCES:
- [Derived] Zoughbie DE, Huddleston D, Watson K, Ding EL. HIV Social-network intervention more effective in older populations in Kenya. BMC Public Health. 2024 Nov 9;24(1):3098. doi: 10.1186/s12889-024-20315-0. PMID 39516844
- [Derived] Hickey MD, Ouma GB, Mattah B, Pederson B, DesLauriers NR, Mohamed P, Obanda J, Odhiambo A, Njoroge B, Otieno L, Zoughbie DE, Ding EL, Fiorella KJ, Bukusi EA, Cohen CR, Geng EH, Salmen CR. The Kanyakla study: Randomized controlled trial of a microclinic social network intervention for promoting engagement and retention in HIV care in rural western Kenya. PLoS One. 2021 Sep 13;16(9):e0255945. doi: 10.1371/journal.pone.0255945. eCollection 2021. PMID 34516557